CLINICAL TRIAL: NCT00587847
Title: Maintenance Alemtuzumab in Refractory Chronic Lymphocytic Leukemia
Brief Title: Campath Maintenance in Chronic Lymphocytic Leukemia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient recruitment.
Sponsor: Northwell Health (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Kanti Rai, MD, Principal Investigator, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05.10.030; Berlex Study# 106.0621 (Other: Berlex)
Record Dates: First submitted 2007-12-21; First posted 2008-01-08 (Estimated); Results first posted 2015-10-15 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-09

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia | interventions — Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Campath maintenance treatment (Other): Single arm, open label trial of Campath on a maintenance schedule for patients who have had a response to prior conventional chemotherapy. Treatments consist of dose escalation (3, 10 and 30mg) during week 1 followed by weekly dosing of Campath at 30 mg once weekly for 7 weeks followed by Campath 30 mg every 2 weeks for 16 weeks followed by Campath 30 mg once every 3 weeks for 24 weeks. Total duration of treatment up to 48 weeks.
  Interventions: Drug: Campath

INTERVENTIONS:
Drug: Campath — Campath 30 mg administered subcutaneously at varying intervals for up to 1 year
  Other Names: Alemtuzumab

SUMMARY:
This is a study designed to test whether giving campath (also known as alemtuzumab) on a maintenance schedule will prolong the time until the patient requires chemotherapy.

DETAILED DESCRIPTION:
This is an open-label, single arm, proof-of-principle study of Campath (also known as alemtuzumab) maintenance therapy administered subcutaneously at varying intervals for up to 1 year. Ongoing prophylactic anti-infectives will be provided. Patients will be assessed for response every 2 months and for quality of life every 3 months while on treatment. Patients achieving a presumptive complete response will receive no further treatment but will be followed for response. Non-responding patients, with confirmed progressing disease following a minimum of 8 doses will be discontinued from treatment and followed for survival. Responding patients or patients with stable disease will undergo confirmatory assessment 2 months following their end-of-treatment assessment. If remission has occurred, patients will be followed off treatment until documented disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in this study is open to patients 18 years of age with confirmed chronic lymphocytic leukemia, a clinical response of stable disease or better to previous treatment, and an Eastern Cooperative Oncology Group performance status of 0-2

Exclusion Criteria:

* Treatment failure in more than 3 prior regimens
* Active secondary malignancy
* Central nervous system involvement with CLL
* History of significant allergic reaction to antibody therapies that required discontinuation of the antibody therapy
* History of HIV positivity
* Hepatitis C virus (HCV) positivity based upon core antigen testing
* Active infection, requiring treatment with antibiotic, antiviral, or antifungal agents
* Pregnancy or lactation
* Other severe, concurrent diseases or mental disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2005-08; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kanti R. Rai, MD, Principal Investigator — Long Island Jewish Medical Center
Locations (1):
- Long Island Jewish Medical Center, New Hyde Park, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was originally designed to recruit 20 patients but only 12 subjects were accrued to the trial before it was stopped due to poor recruitment. Subjects were entered between August 2005 and July 2007. All subjects had Chronic Lymphocytic Leukemia that was previously treated with chemotherapy.
Groups:
- Single Arm, Open Label Trial.: single arm, open label trial using Campath 30 mg administered subcutaneously at varying intervals for up to 1 year.
Period: Overall Study
Arm/Group | Single Arm, Open Label Trial.
Started | 12
Completed | 5
Not Completed | 7
Not completed — Lack of Efficacy | 5
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Population: This was a pilot study with enrollment goal of 20 based on our patient population with potential to meet inclusion criteria. This goal was not met due to patient preferance for no further treatment which is standard of care.
Arm/Group | Single Arm, Open Label Trial.
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression (Months)
Description: Time to progression calculated as the period, in months, between the date of the first dose of alemtuzumab and the first date of documented disease progression (NCI 1996 criteria) or death. Duration of response of all other participants who did not progress nor expire, had their event times calculated at the last date of follow-up.
Time Frame: Every 8 weeks
Population: All patients who were entered on study were analyzed according to NCI Working Group Response Criteria for CLL. Adverse events were graded on a scale of 1 to 4, where possible, according to the NCI Common Toxicity Criteria, Version 2.0.
Measure: Mean (Full Range); unit: months
Arm/Group | Single Arm, Open Label Trial.
Number analyzed (Participants) | 12
months | 10 [3 to 22]

2. Secondary Outcome: Rate of Infections
Description: Number of participants who developed clinical or laboratory evidence of infection.
Time Frame: Weekly then every 2 weeks then every 3 weeks
Population: All participants who received at least one dose of alemtuzumab were analyzed for safety.
Measure: Number; unit: participants
Groups:
- All Participants: All participants were included in the safety analysis.
Arm/Group | All Participants
Number analyzed (Participants) | 12
participants | 2

ADVERSE EVENTS:
Arm/Group | Single Arm, Open Label Trial.
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 5/12
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm, Open Label Trial. (N=12)
Injection Site reaction (General disorders) | 2 (2) — mild, grade 1 injection site reaction seen in 2 participants
Lung infection (Infections and infestations) | 1 (1) — Grade 2 pneumonia
Autoimmune disorder (Immune system disorders) | 2 (2) — Grade 3 Immune Thrombocytopenia (ITP)

LIMITATIONS AND CAVEATS:
Trial was terminated early due to poor accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No